CLINICAL TRIAL: NCT00188253
Title: Positron Emission Tomography Scanning and Epstein-Barr Virus DNA Levels in the Staging and Follow-up of Nasopharyngeal Carcinoma.
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 04-0264-C
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; PET scan; MRI; EBV virus
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The standard treatment for nasopharyngeal cancer involves either radiation alone or radiation plus chemotherapy. Before the start of treatment,patients require an imaging scan to assess the extent of disease. The most commonly used test is a magnetic resonance imaging (MRI) scan.

The goal of the study is to examine the value of a new imaging technology that has recently become available at the University Health Network Hospitals called Positron Emission Tomography scanning (PET). PET scanning involves the injecting a small amount of a drug through a vein in the arm called 18-fluorodeoxyglucose (18FDG). This drug is special in that it is radioactive and will be detected by the PET machine. Cancer cells are believed to be more active than normal cells and have a high rate of metabolism. Therefore, cancer cells are thought to take up glucose (a kind of sugar) faster than normal cells in the body. Because 18FDG is a modified type of glucose, it is also taken up by cancer cells. Special imaging cameras will be able to visualize the areas of uptake and reveal sites of cancer involvement. The main goal of this study is to evaluate whteher the scan is able to detect the presence of nasopharyngeal carcinoma (NPC) both before and after treatment and to specifically compare it to findings on magnetic resonance imaging scans (MRI).

In addition to doing the PET scans, we are asking patients to have blood samples drawn throughout their treatment and follow-up, for a research test called Epstein Barr virus (EBV) DNA levels. The Epstein Barr virus is thought to have a role in the development of nasopharyngeal cancer, and many patients with nasopharyngeal carcinoma are found to have high levels of EBV DNA levels in their blood. The second goal of this study is to evaluate whether changes in EBV DNA levels are associated with the treatment and the disease course in nasopharyngeal cancer, and whether they help to predict any changes in the cancer. This part of the study involves the sampling of a small amount of venous blood at a time prior to the beginning of therapy and at regular intervals following treatment.

DETAILED DESCRIPTION:
1. Patients with nasopharyngeal carcinoma are staged according to the 2002 American Joint Committee on Cancer (AJCC) criteria. MRI is the imaging modality of choice for staging and follow-up of nasopharyngeal carcinoma. The goal is to conduct a pilot study to compare the staging findings on MRI with those on PET scanning in both pre- and post-therapy patients. The end point is to document the degree of concordance between the two modalities with respect to the anatomic location and volume of disease at the time of initial staging and on follow up and to determine how any differences observed may alter staging and management including radiation planning. We hypothesize that PET scanning will be able to detect recurrence and residual disease within the radiated tissue earlier than MRI.
2. Nasopharyngeal carcinoma is associated with elevated titers of Epstein Barr virus (EBV) cell free, plasma DNA. Fluctuation i.e. - elevation in EBV DNA levels following therapy may serve as a potential marker for recurrent or residual disease. We believe that a change in EBV DNA titer precedes changes on conventional MRI and possibly PET scans in patients with recurrent disease. We also predict, that due to its sensitivity, that EBV titer levels will be more sensitive in the evaluation of tumor response to therapy, as well predicting tumor recurrence. The second goal is to conduct a trial to compare the sensitivity of MRI, PET and EBV titers in the assessment of recurrent disease.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients with histologically diagnosed nasopharyngeal carcinoma presenting to the University Health Network for which a course of curative radiation therapy +/- chemotherapy is planned.

2. Patient is able to provide informed consent and is willing to adhere to the study protocol.

Exclusion Criteria:

- 1. Patients with metastatic disease. 2. Lactating or pregnant females. 3. Medical or psychological conditions such as claustrophobia, etc., that in the opinion of the referring MD or study investigator, would make the patient unable to tolerate the study procedures.

4. Presence of a second malignancy or a history of another malignancy active within the last 5 years, with the exception of non-head and neck, non-melanomatous cutaneous malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically diagnosed nasopharyngeal carcinoma presenting to the University Health Network for which a course of curative radiation therapy +/- chemotherapy is planned.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2005-03; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Yu, MD, Principal Investigator — University Health Network, University of Toronto
Locations (1):
- Princess Margaret Hospital, University Health Network, Toronto, Ontario, Canada